CLINICAL TRIAL: NCT06276569
Title: A Single-center, Randomized, Controlled, Study Evaluating the Efficacy and Safety of Sivelestat Sodium in Preventing Postoperative Acute Lung Injury or Acute Respiratory Distress Syndrome Following Cardiac Surgery
Brief Title: Efficacy and Safety of Sivelestat in Preventing Postoperative Acute Lung Injury or Acute Respiratory Distress Syndrome After Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-LCYJ-MS-26
Record Dates: First submitted 2024-01-31; First posted 2024-02-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases | interventions — sivelestat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sivelestat group (Experimental): sivelestat was dissolved in 0.9% sodium chloride injection and diluted with 50ml of the same solution to achieve a dose of 4.8mg/kg/day; this mixture was then placed in a sealed package and administered intravenously at a rate of 0.2 mg/kg/h for seven consecutive days.
  Interventions: Drug: Sivelestat
- placebo comparator (Placebo Comparator): received an equivalent volume (50ml) of saline continuously administered intravenously at a rate of 0.2 mg/kg/hour.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Sivelestat — (1)Experimental group: Received intravenous sivelestat sodium admission to the ICU. Sivelestat sodium was dissolved in 0.9% sodium chloride injection and a one-day dose (4.8mg/kg) was diluted in 50ml of 0.9% sodium chloride injection, which was then sealed for continuous intravenous administration at a rate of 0.2 mg/kg/h for seven consecutive days.
  Arms: sivelestat group
Other: placebo — 2)Control group: Receiving the same dose of placebo, 50 ml of saline, were administered intravenously at a rate of 0.2 mg/kg throughout the treatment period without any discernible impact on patient's regular treatment regimen.
  Arms: placebo comparator

SUMMARY:
The aim of this study is to assess the effectiveness and safety of sivelestat sodium in preventing acute lung injury and/or acute respiratory distress syndrome (ALI/ARDS) following cardiac surgery, with the objective of providing evidence-based support for its clinical application.

DETAILED DESCRIPTION:
This study is being performed as a randomized, placebo-controlled trial conducted in 442 patients who met the inclusion and exclusion criteria and were scheduled for elective cardiac surgery. Following informed consent, patients were randomly assigned to either the experimental group or the control group, with the study drug administered after transfer to the ICU post-surgery. In the experimental group, sivelestat was dissolved in 0.9% sodium chloride injection and diluted with 50ml of the same solution to achieve a dose of 4.8mg/kg/day; this mixture was then placed in a sealed package and administered intravenously at a rate of 0.2 mg/kg/h for seven consecutive days. The control group received an equivalent volume (50ml) of saline continuously administered intravenously at a rate of 0.2 mg/kg/hour. Demographic and clinical information, including admission diagnosis, underlying diseases, medical history, surgical history, details of the surgical procedure, postoperative complications, and in-hospital outcomes were collected from all participants. The primary outcome is the incidence of postoperative ARDS. Secondary outcome measures include data collection on the following parameters: elevated inflammatory response indices (WBC>20×109/L; IL-6>301.88mg/ml; CRP>49.76mg/L; PCT>2.18ng/ml) on postoperative days 1, 3, 5, and 7; APACHE II score; Murray lung injury score; incidence of severe pneumonia; mechanical ventilation-free rate at day 28; mortality rates at both day 28 and day 90. Adverse events such as liver injury, leukopenia, and thrombocytopenia resulting from sivelestat treatment were also monitored. Additionally,during the follow-up period, mortality within a 90-day period will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 50 and 80 years old.
2. Both sexes.
3. Patients undergoing elective cardiac surgery;informed consent.

Exclusion Criteria:

1. Patients undergoing emergency surgery.
2. Patients undergoing deep hypothermic circulatory arrest surgery;.
3. Patients with liver and kidney dysfunction (Child-Pugh class B or C, estimated glomerular filtration rate <35 mL/min/1.73 m2).
4. Patients with abnormal baseline inflammatory markers [interleukin-6 (IL6) >10 pg/mL, procalcitonin (PCT) >0.5 ng/mL, C-reactive protein (CRP) >10 mg/L].
5. Patients diagnosed with inflammatory immune disease, infectious disease, or oncological disease; patients receiving other medications that inhibit neutrophil elastase (e.g., ulinastatin, alpha 1-antiprotease).
6. Patients allergic to or intolerant to sodium sivelestat.
7. Pregnant.
8. Patients with prognostic mortality on the European System for Cardiac Surgery Risk Evaluation II (EuroSCORE II) >3% were randomly assigned to either the treatment group or the control group based on the inclusion and exclusion criteria.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2024-02-18 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Oxygenation index | postoperative day 1, 3, 5 and 7
  SpO2 /FIO2
Inflammatory index | postoperative day 1, 3, 5 and 7
  WBC[×109/L], Neutrophil[NEU,%], Interleukin(IL)-1β[pg/mL], IL-6[pg/mL], IL-8[pg/mL], TNF-α[pg/mL], CRP[mg/L], PCT[ng/mL], neutrophil elastase[NE,ng/mL] and myeloperoxidase[MPO, ng/ml]
Myocardial injury marker | postoperative day 1, 3, 5 and 7
  myoglobin[Myo, ng/ml], CK-MB[ng/ml], hs-cTnI[ng/ml]
Acute physiology and chronic health evaluation(APACHE II) socre | postoperative day 1, 3, 5 and 7
  Interpretation of APACHE II : minimum 0 and maximum 71; increasing score is associated with an increasing risk of hospital death. acute physiology score, chronic health status score, and age adjustment score
Murray socre | postoperative day 1, 3, 5 and 7
  Interpretation of Murray socre : the Murray Lung Injury Score, a clinical assessment tool for evaluating the severity of acute lung injury. The score ranges from 0 to 4, with higher scores indicating worse pulmonary function and more severe lung injury.
ICU time | postoperative 28 days
  Time to stay in the intensive care unit
In-hospital time | postoperative 28 days
  All time during hospitalization
30-day all-cause mortality | postoperative 30 dayS
  Proportion of deaths caused by various reasons within a certain period of time (30 days) compared to the total number of people in a certain group
90-day all-cause mortality | postoperative 90 days
  Proportion of deaths caused by various reasons within a certain period of time (90 days) compared to the total number of people in a certain group

CONTACTS AND LOCATIONS:
Overall Officials: Tuo Pan, MD, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, China

IPD SHARING:
Plan to Share IPD: No